CLINICAL TRIAL: NCT06825052
Title: Effects of Deloading Periods in Resistance Training on Muscular Strength and Hypertrophy in Untrained Young Individuals: A Randomized Controlled Trial
Brief Title: Effects of Deloading Periods in Resistance Training on Muscular Strength and Hypertrophy
Acronym: DPRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Zarife Pancar, PhD, Assistant Professor,, University of Gaziantep
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: GAUN-SBF-PANCAR-02; OFS (Registry Identifier: 7a55420f9c0843838b7da349ba26195f)
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Muscle Hypertrophy in Healthy Young Men
Keywords: Muscle hypertrophy; muscle strength; resistance training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This study utilizes a crossover within-subject design, where each participant's limbs were assigned to two different training conditions:
  Deload Training Condition: Training volume and frequency were reduced for one week every four weeks.
  Continuous Training Condition: Training continued without volume reduction. Each participant performed unilateral leg extension and dumbbell biceps curl exercises twice per week for 8 weeks. One limb was assigned to the deload condition, while the other was assigned to the continuous training condition.
  This within-subject design was chosen to minimize inter-individual variability and enhance statistical power. Muscle hypertrophy and strength were assessed before and after the intervention using B-mode ultrasound and 10-repetition maximum (10RM) testing, respectively.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study utilized a double-blind (participant and outcomes assessor) design to minimize bias in the evaluation of muscle hypertrophy and strength.
  Participants were unaware of which limb was assigned to the deload or continuous training condition to prevent psychological or behavioral influences on training performance.
  The outcomes assessor conducting muscle thickness measurements (using B-mode ultrasound) and strength assessments (10RM test) was blinded to the condition assignments to ensure unbiased data collection.
  The researchers responsible for training supervision were aware of the limb assignments but did not participate in the measurement or data analysis process.
  This blinding method was implemented to enhance the validity of the study and reduce potential bias in both subjective and objective outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deload Training (Experimental): Participants in this group followed an 8-week resistance training program with deloading periods every four weeks. During these deload weeks, training volume and intensity were reduced to facilitate recovery while maintaining training adaptations.
  Interventions: Behavioral: Resistance Training with Deloading Periods
- Continuous Training (Active Comparator): Participants in this group followed an 8-week continuous resistance training program with no reductions in training volume or intensity. This group served as a comparison to assess the effects of deloading periods on muscle hypertrophy and strength.
  Interventions: Behavioral: Continuous Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training with Deloading Periods — Participants performed an 8-week unilateral resistance training program in which training volume and intensity were reduced during weeks 4 and 8 to facilitate recovery and adaptation.
  Arms: Deload Training
Behavioral: Continuous Resistance Training — Participants followed an 8-week unilateral resistance training program without any deloading periods. Training volume and intensity remained consistent throughout the study.
  Arms: Continuous Training

SUMMARY:
This study investigates the effects of deloading periods (short breaks or reductions in training volume) in a 8-week resistance training program on muscle strength and hypertrophy in young, untrained individuals.

Participants were randomly assigned to two training conditions:

Deload Training Group: Reduced training volume for one week every four weeks. Continuous Training Group: Regular training without reductions. Muscle thickness was measured using ultrasound, and muscle strength was evaluated through a 10-repetition maximum (10RM) test before and after the intervention.

The findings showed that both training strategies led to significant increases in muscle strength and size, with no major differences between groups. This suggests that incorporating deloading periods does not negatively impact muscle development and may serve as an effective alternative for individuals with time constraints or minor injuries.

This study was conducted at Gaziantep University, Faculty of Sports Sciences, with approval from the university's ethics committee.

DETAILED DESCRIPTION:
This study examines the effects of deloading periods (planned reductions in training volume and frequency) within an 8-week resistance training program on muscle hypertrophy and strength in untrained young individuals.

The study utilized a randomized within-subject design, where each participant's limbs were assigned to one of two conditions:

Deload Training Condition: Training volume and frequency were reduced during Weeks 4 and 8 to allow for recovery.

Continuous Training Condition: No reductions in training volume were applied. The resistance training program included unilateral leg extension and unilateral dumbbell biceps curl exercises performed twice per week. The training intensity was adjusted to ensure participants reached voluntary muscular failure within the 8-12 repetition range.

Assessments & Measurements:

Muscle Hypertrophy: Measured using B-mode ultrasound at different quadriceps and biceps locations.

Muscle Strength: Evaluated through 10-repetition maximum (10RM) testing before and after the intervention.

Statistical Analysis: A 2-way repeated-measures ANOVA was used to compare training conditions, with effect sizes analyzed to determine the significance of adaptations.

The study was approved by the Gaziantep University Health and Sports Sciences Ethics Committee and conducted in accordance with the Declaration of Helsinki guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, untrained individuals (no prior structured resistance training experience for at least 6 months).
* Aged between 18-25 years old.
* No current or recent musculoskeletal injuries affecting exercise performance.
* No diagnosed medical conditions that could interfere with resistance training.
* Willing to participate in an 8-week structured resistance training program.
* No use of performance-enhancing drugs, anabolic steroids, or other muscle-growth supplements.

Exclusion Criteria:

* Individuals with prior resistance training experience within the last 6 months.
* Any current or past musculoskeletal injuries or conditions affecting the lower or upper limbs.
* Any diagnosed metabolic, cardiovascular, or neurological disorders that could affect physical performance.
* Individuals currently taking medications that affect muscle function or recovery.
* Pregnant or breastfeeding individuals.
* Failure to comply with the study protocol (e.g., missing more than 2 training sessions).

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants were eligible to participate in the study. Gender identity was not a restriction, but biological sex was considered for eligibility.
Enrollment: 19 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Muscular Strength | Baseline and after 8 weeks
  Changes in muscle strength will be assessed using 10-repetition maximum (10RM) testing before and after the intervention. Strength assessments will be conducted for both the quadriceps (leg extension) and biceps brachii (dumbbell curl).

SECONDARY OUTCOMES:
Muscle Hypertrophy | Baseline and after 8 weeks
  Changes in muscle thickness will be measured using B-mode ultrasound imaging. Measurements will be taken at multiple anatomical points on the quadriceps and biceps brachii muscles before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Zarife Pancar Assistant Professor,, PhD, Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep University, Faculty of Sport Sciences, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with other researchers upon reasonable request. Data will be available after study completion and publication, following ethical approval and data-sharing agreements. Researchers interested in accessing the data may contact the corresponding author.
Supporting Information: Study Protocol, CSR
Time Frame: De-identified individual participant data (IPD), along with the study protocol and statistical analysis plan, will be made available upon request after study completion and publication. Researchers interested in accessing the data should contact the corresponding author. Data will be shared under a data-sharing agreement to ensure compliance with ethical and privacy guidelines.
Access Criteria: De-identified individual participant data (IPD) and supporting documents, including the study protocol and statistical analysis plan, will be available upon reasonable request for research purposes. Access will be granted to qualified researchers affiliated with academic or research institutions. Researchers must submit a data-sharing request, including a brief study proposal outlining their intended use of the data. All data-sharing requests will be reviewed by the study team, and approved researchers must sign a data-sharing agreement to ensure compliance with ethical and privacy guidelines. Data will be shared in a secure format via institutional data-sharing platforms or encrypted file transfer.
URL: https://osf.io/6cgpt/?view_only=7a55420f9c0843838b7da349ba26195f